CLINICAL TRIAL: NCT01905631
Title: A 3-Day Investigator Blinded, Randomized Study Evaluating Aurstat Anti-Itch Hydrogel Versus Control in the Treatment of Atopic Dermatitis Associated Pruritus
Brief Title: Blinded, Randomized Study Evaluating Aurstat Versus Control in the Treatment of Atopic Dermatitis Associated Pruritus
Acronym: AUR0613
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Center for Clinical and Cosmetic Research (Other)
Collaborators: Onset Dermatologics, Inc. (Unknown)
Responsible Party: Principal Investigator, Mark Steven Nestor, M.D., Ph.D., Director, The Center for Clinical and Cosmetic Research
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: AUR0613
Record Dates: First submitted 2013-07-19; First posted 2013-07-23 (Estimated); Results first posted 2022-10-24 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Pruritus; Atopic Dermatitis
Keywords: Pruritus; Atopic Dermatitis
MeSH Terms: conditions — Pruritus; Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Untreated Control Group (No Intervention): Subjects will apply nothing for the entire three days of the trial. Subjects will also fill out a study diary assessing adverse events or other events they experience during the trial.
- Treatment Group (Aurstat) (Active Comparator): Subjects will apply Aurstat Anti-Itch Hydrogel 2 times daily or as needed for up to three days to reduce itching. Subjects will also fill out a study diary assessing adverse events or other events they experience during the trial.
  Interventions: Drug: Aurstat Anti-Itch Hydrogel (Aurstat)

INTERVENTIONS:
Drug: Aurstat Anti-Itch Hydrogel (Aurstat) — Subjects will apply Aurstat Anti-Itch Hydrogel 2 times daily or as needed for up to three days to reduce itching. Subjects will also fill out a study diary assessing adverse events or other events they experience during the trial.
  Arms: Treatment Group (Aurstat)

SUMMARY:
To demonstrate the ability of Aurstat to reduce pruritus in subjects with mild to moderate atopic dermatitis. Efficacy results will be based on subject assessment, IGA, and photographic evidence based on ordinal scales for tolerability.

DETAILED DESCRIPTION:
This 3-day study will enroll subjects with mild to moderate atopic dermatitis, as defined by the Hanifin criteria.

All subjects will be screened for study enrollment at the baseline visit. Those meeting inclusion/exclusion criteria will be fully consented (or assented) using an IRB-approved ICF. Subjects will then be randomized to either the treatment or control study arm. Those in the treatment arm will be instructed on product application technique and study instructions at baseline. Subjects will apply Aurstat BID, or as needed, to determine frequency of use as a surrogate marker for duration of therapy effect to affected, qualifying atopic dermatitis lesions.

The investigator will assess treatment response using an ordinal scale for tolerability and an IGA scale for disease severity ratings. Subjects will assess treatment response using a VAS to rate pruritus and an ordinal scale to assess tolerability. Photography assessments will be obtained. All adverse events will be captured.

ELIGIBILITY:
Inclusion Criteria:

Patients who meet all of the following criteria are eligible for this study.

1. Subjects must be diagnosed by the investigator as meeting the criteria for mild to moderate atopic dermatitis, as defined by the Hanifin criteria.
2. Subjects must score a minimum of 2 on the itch severity scale.
3. Subjects may not apply other topical products (including moisturizers) to the affected lesions, other than study treatments, for a minimum of 24 hours prior to study initiation and for the duration of the study.
4. No other oral or topical treatments for atopic dermatitis are allowed during the study.
5. Subjects on asthma or allergy medications must continue taking these prescription or OTC products without change during the study.
6. Anti-inflammatory oral medications or oral antihistamines not used at cannot be added during the study or taken on an intermittent basis.
7. Subjects must be 12-75 years of age with no known medical conditions that, in the investigator's opinion, may interfere with study participation, except mild to moderate atopic dermatitis.
8. Women of childbearing potential must be willing to use a form of birth control during the study. For the purpose of this study, the following are considered acceptable methods of birth control: oral contraceptives, Norplant, Depo-Provera, double barrier methods (e.g., condom and spermicide), and abstinence.

Exclusion Criteria:

Patients who meet any of the following criteria are not eligible for this study.

1. Any dermatological disorder, which in the investigator's opinion, may interfere with the accurate evaluation of the subject's response to the study formulation.
2. Subjects who have demonstrated a previous hypersensitivity reaction to any of the ingredients of the study product.
3. Concurrent therapy with any medication either topical or oral that might interfere with the investigator and/or subject assessments of atopic dermatitis or study product irritancy, based on the opinion of the investigator.
4. Subjects who have used a topical corticosteroid within 2 weeks of study enrollment.
5. Subjects who are on oral corticosteroids within 4 weeks of study enrollment, inhaled corticosteroids are allowed if used at baseline and used on a routine basis. Intermittent inhaled corticosteroids are prohibited.
6. Subjects who use an indoor tanning booth.
7. Subjects who are pregnant, breast feeding or planning a pregnancy.
8. Subjects with clinically significant unstable medical disorders.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-07; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Berman, MD, PhD, Principal Investigator — Center for Clinical and Cosmetic Research; Mark S. Nestor, MD, PhD, Principal Investigator — Center for Clinical and Cosmetic Research
Locations (1):
- Center for Clinical and Cosmetic Research, Aventura, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Untreated Control Group | Treatment Group (Aurstat)
Started | 10 | 20
Completed | 10 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Untreated Control Group | Treatment Group (Aurstat) | Total
Number analyzed (Participants) | 10 | 20 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 18 | 28
  >=65 years | 0 | 2 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.2 (5.3) | 51.5 (6.8) | 47.1 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 22
  Male | 0 | 8 | 8
Region of Enrollment [Number; unit: participants]
  United States | 10 | 20 | 30

OUTCOME MEASURES:

1. Primary Outcome: Reduction of Itching in AD
Description: The ability of Aurstat to reduce itching in those diagnosed with Atopic Dermatitis aged 12-75 years of age.
  Visual analog score (VAS assessment)- the VAS itch score was defined as the number of millimeters from the left side of a line (154 mm in length) that indicates their level of itching (0 mm (no itching)-154 mm (most itching)).
Time Frame: 3-days
Population: Itch score
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Untreated Control Group | Treatment Group (Aurstat)
Number analyzed (Participants) | 10 | 20
score on a scale | 1.70 (0.483) | 1.55 (0.826)

ADVERSE EVENTS:
Time Frame: 3 days
Description: Patients in the placebo group were not at risk for serious adverse effects.
Arm/Group | Untreated Control Group | Treatment Group (Aurstat)
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/20
Other Adverse Events (participants affected / at risk) | 0/10 | 1/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Untreated Control Group (N=10) | Treatment Group (Aurstat) (N=20)
Facial dryness (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Facial dryness associated with use of IP. Problem resolved with application of gel to face and was noted as a protocol deviation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes